CLINICAL TRIAL: NCT05277493
Title: A Registry of Chinese AL Amyloidosis Patients Treated With Subcutaneous or Intravenous Daratumumab
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AL amyloidosis registry
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: AL Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this protocol is to generate a registry of Chinese patients with AL amyloidosis treated with subcutaneous/intravenous daratumumab alone or subcutaneous/intravenous daratumumab combined with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* newly diagnosed or refractory/relapsed AL amyloidosis
* treated with subcutaneous/intravenous daratumumab alone or subcutaneous/intravenous daratumumab combined with chemotherapy

Exclusion Criteria:

* co-diagnosis of multiple myeloma or Waldenström's macroglobulinemia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled in this registry pending on expressing an informed consent of the use of their data for research purposes
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Hematologic complete response at 3 months | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China